CLINICAL TRIAL: NCT05773365
Title: Evaluation of Analgesic Effect of Added Local Infiltration to Pericapsular Nerve Group Block in Traumatic Hip Surgery
Brief Title: PENG Block Plus Local Infiltration Compared to PENG Block Alone in Hip Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5177
Record Dates: First submitted 2023-03-06; First posted 2023-03-17 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Pain; Hip Fractures; Postoperative Pain; Postoperative Analgesia
MeSH Terms: conditions — Pain; Hip Fractures; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pericapsular Nerve Group Block plus local infiltration (Experimental): Group A (study group) will receive both PENG block and local infiltration at the end of the surgery.
  Spinal anaesthesia will be administered to the patient using 7.5-12.5 mg heavy 0.5% bupivacaine at L3-L5 lumbar spine using 25 G spinal needle.
  If spinal anaesthesia is contraindicated or failed, patients will have general anaesthetics.
  General anaesthesia will be induced with 2-3 mcg/kg fentanyl, Propofol 1-2 mg/kg titrated to effect, and muscle relaxant if required.
  PENG block will be administered according to the description by injecting 20 ml of 0.25% bupivacaine below the psoas tendon.
  A 20 ml of 0.25% bupivacaine will be infiltrated by the surgeons to the tissues at the end of the surgery.
  Interventions: Other: PENG block with or without local anaesthetic infiltration
- Pericapsular Nerve Group Block (Active Comparator): In Group B, only PENG block will be administered in this arm
  Interventions: Other: PENG block with or without local anaesthetic infiltration

INTERVENTIONS:
Other: PENG block with or without local anaesthetic infiltration — As mentioned.

SUMMARY:
Summary:

Pain control after hip surgery is quite important for patients' recovery. Many regional techniques are available with the focus on motor sparing block to speed patient recovery.

The investigators will compare pericapsular nerve group (PENG) block in addition to local skin infiltration to PENG block alone. The study population will be included for patient traumatic hip surgery. The study population will be divided into group. First group will receive PENG block and local anaesthetics infiltration and second group will receive PENG block.

Our primary outcome is to compare numeric rating scale (NRS) between studied groups, and morphine requirements in the first 24 hours as a secondary outcome.

DETAILED DESCRIPTION:
Aim of the study:

The aim of the study is to improve quality of patient's post-operative recovery after hip surgery.

Study objectives:

To compare Patient numeric rating scale (NRS) scores after hip surgery for patients receiving PENG block and local skin infiltration

Study question:

Will PENG block and local infiltration provide significant analgesia for hip surgery than PENG block alone?

Null Hypothesis:

Local infiltration addition to PENG block will not provide significant analgesia to PENG block alone.

Alternative hypothesis:

Local infiltration addition to PENG block will provide significant superior analgesia to PENG alone.

Study Design:

Single blinded randomized clinical trial. Ethical approval will be obtained from Suez Canal University. Patients' enrolment will be obtained preoperatively. Patients' demographic data will be recorded (age, weight, BMI, and gender).

An informed consent will be obtained during enrolment explaining the aim of the study and complication of the techniques. Patient will have the right to withdraw from the study at any time.

Patients will be randomly allocated to either of the studied group through the following method:

Randomization of the patients meeting the inclusion criteria will be achieved by a computer-generated random sequence, and this sequence will be concealed in sealed numbered envelopes, labelled Group A (study group) carry the label Group B (control group).

Methods:

Group A (study group) will receive both PENG block and local infiltration at the end of the surgery. Group B (control group) will receive PENG block without local infiltration.

Spinal anaesthesia will be administered to the patient using 10-12.5 mg heavy 0.5% bupivacaine at L3-L5 lumbar spine using 25 G spinal needle.

If spinal anaesthesia is contraindicated or failed, patients will have general anaesthetics.

General anaesthesia will be induced with 1-2 mcg/kg fentanyl, propofol 1-2 mg/kg, and appropriate muscle relaxant.

Block will be administered for trauma patients PENG block will be administered as following:

A curvilinear US sound probe will be placed in a transverse plane over anterior superior iliac spine and rotated 45 degrees anticlockwise till identifying femoral vessels, iliopubic eminence, iliopsoas muscle tendon in the view. A 100 mm echogenic needles (SonoPlex STIM, Germany) will be advanced from lateral to medial and injecting 20 ml of 0.25% bupivacaine below the psoas tendon.

A 20 ml of 0.25% bupivacaine will be infiltrated by the surgeons to the tissues at the end of the surgery.

Pain management:

All patients will receive 1g of paracetamol, 30 mg Ketorolac, and 8 mg Dexamethasone after spinal anaesthesia.

Postoperatively 1g of paracetamol four times a day, ketorolac 30 mg twice a day for 48 hours. Intravenous morphine 2 mg every 10 minutes will be given to the patient if NRS score ≥ 4 till pain is controlled as rescue analgesics.

Morphine requirement will be assessed in recovery and then every 6 hours, in the first 24 hours after surgery. If the pain score > 4, patient will get 2 mg IV morphine. Pain will be reassessed after 10 minutes for further analgesia requirement.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anaesthesiology (ASA) 1-3
2. Traumatic hip surgeries (total hip arthroplasty, hemiarthroplasty, Dynamic hip screw).

Exclusion Criteria:

1. Patient with cognitive impairment.
2. Patient weight < 50 kg.
3. Allergy to medications used.
4. Chronic kidney disease. (serum creatinine > 2.5 mg/dl).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain scores | 24 hours
  The difference in patient numeric rating scale (NRS). 11 points scale, where 0 means no pain and 10 is worst possible pain. The higher pain scores means worse outcome between both groups.

SECONDARY OUTCOMES:
Morphine requirement | 24 hours
  Postoperative morphine requirement

CONTACTS AND LOCATIONS:
Overall Officials: Eslam Albayadi, Principal Investigator — Suez Canal University, Ring Road, Ismailia, Egypt
Locations (1):
- Suez Canal University Hospital, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young AC, Buvanendran A. Pain management for total hip arthroplasty. J Surg Orthop Adv. 2014 Spring;23(1):13-21. doi: 10.3113/jsoa.2014.0013. PMID 24641893
- [Background] Tran DQ, Salinas FV, Benzon HT, Neal JM. Lower extremity regional anesthesia: essentials of our current understanding. Reg Anesth Pain Med. 2019 Jan 11:rapm-2018-000019. doi: 10.1136/rapm-2018-000019. Online ahead of print. PMID 30635506
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Pascarella G, Costa F, Del Buono R, Pulitano R, Strumia A, Piliego C, De Quattro E, Cataldo R, Agro FE, Carassiti M; collaborators. Impact of the pericapsular nerve group (PENG) block on postoperative analgesia and functional recovery following total hip arthroplasty: a randomised, observer-masked, controlled trial. Anaesthesia. 2021 Nov;76(11):1492-1498. doi: 10.1111/anae.15536. Epub 2021 Jul 1. PMID 34196965
- [Background] Lin DY, Brown B, Morrison C, Fraser NS, Chooi CSL, Cehic MG, McLeod DH, Henningsen MD, Sladojevic N, Kroon HM, Jaarsma RL. The Pericapsular Nerve Group (PENG) block combined with Local Infiltration Analgesia (LIA) compared to placebo and LIA in hip arthroplasty surgery: a multi-center double-blinded randomized-controlled trial. BMC Anesthesiol. 2022 Aug 6;22(1):252. doi: 10.1186/s12871-022-01787-2. PMID 35933328